CLINICAL TRIAL: NCT03804086
Title: Clinical and Radiographic Evaluation of Advanced Platelet Rich Fibrin Combined With Nano-crystalline Hydroxyapatite Bone Substitute for Management of Mandibular Molar Grade II Furcation Defects
Brief Title: Evaluation of Advanced PRF Combined With Nano-crystalline Hydroxyapatite for Management of Grade II Furcation Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadeer Ashraf Hassan Roushdy (Other)
Responsible Party: Sponsor-Investigator, Hadeer Ashraf Hassan Roushdy, Dentist, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: perio2019
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Advanced PRF (A-PRF) + nano-crystalline hydroxyapatite bone substitute combined with open flap debridement (OFD).
  Interventions: Procedure: Advanced PRF (A-PRF) + nano-crystalline hydroxyapatite bone substitute combined with open flap debridement
- Control Group (Active Comparator): Open flap debridement alone.
  Interventions: Procedure: Open flap debridement

INTERVENTIONS:
Procedure: Advanced PRF (A-PRF) + nano-crystalline hydroxyapatite bone substitute combined with open flap debridement — will treated with OFD +A- PRF+ nano-crystalline hydroxyapatite bone substitute,10 mL of blood will be drawn from only patient assigned to the intervention group by vein puncture of the antecubital vein and is collected in sterile glass test tube, without any anticoagulant.
  * The blood will be quickly collected, and the tube will immediately centrifuge at 1500 rpm for14 min at room temperature.
  * After centrifugation, the A-PRF clot will be removed from the tube using sterile tweezers and placed on sterile woven gauze. Membrane will prepared by compressing clots between two pieces of woven gauze.
  Arms: Test Group
Procedure: Open flap debridement — a periodontal access flap will be initiated by intrasulcular incisions on the buccal and lingual aspects. The incisions will be carried as far interproximally as possible to preserve the entire Interdental papillae and to achieve primary wound closure.
  Arms: Control Group

SUMMARY:
this study is to evaluate the use of advanced platelet rich fibrin (A-PRF) + nano-crystalline hydroxyapatite bone substitute combined with open flap debridement (OPD) versus open flap debridement alone in the management of mandibular molar grade II defects.

In the management of mandibular molar grade II furcation defects, no difference exists in gain of horizontal clinical attachment level between the use of advanced platelet rich fibrin (A-PRF) + with nano-crystalline hydroxyapatite bone substitute combined with open flap debridement (OPD) and open flap debridement (OPD) alone .

ELIGIBILITY:
Inclusion Criteria:

Patient-related criteria:

* Systemically healthy patients.
* Compliance with oral hygiene instructions and the maintenance program provided.
* Accepts the 6 months follow-up period.
* Provide informed consent.

Teeth related criteria:

* Mature permanent tooth.
* Asymptomatic mandibular molar with buccal Glickman class II furcation involvement.
* Probing depth (PD) ≥ 5 mm and vertical PD ≥ 3 mm after Phase I therapy (scaling and root planing).
* Presence of radiolucency in the furcation area on an intra-oral periapical radiograph

Exclusion Criteria:

Patient-related criteria:

* Patients taking drugs known to interfere with periodontal wound healing in the last six months.
* Pregnant or nursing women.
* Smokers.
* Uncooperative patients.

Teeth related criteria:

* Teeth with interproximal supra-bony or intrabony defects.
* Teeth with gingival recession.
* Teeth with grade II or III mobility.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Relative Vertical Clinical Attachment Level (RVCAL) | 6 months
  relative vertical clinical attachment level (RVCAL) along with gingival marginal level (GML) will be measured from the apical level of customized acrylic stents with grooves to ensure a reproducible placement of a periodontal probe

SECONDARY OUTCOMES:
Relative Horizontal Clinical Attachment Level (PHCAL) | 6 months
  relative vertical clinical attachment level (RVCAL) along with gingival marginal level (GML) will be measured from the apical level of customized acrylic stents with grooves to ensure a reproducible placement of a periodontal probe
Probing Depth (PD) | 6 months
  Probing depth measured from the gingival margin to the base of the pocket.
Gingival margin Level (GML) | 6 months
  • Williams graduated probe will be used for vertical measurement and gingival margin level and Nabers probe for horizontal measurements.

IPD SHARING:
Plan to Share IPD: Undecided